CLINICAL TRIAL: NCT00605618
Title: A Phase I/II Multiple Ascending Dose Study of BMS-777607 in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: Multiple Ascending Dose Study of BMS-777607 in Subjects With Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA192-002
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2009-08

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — N-(4-(2-amino-3-chloropyridin-4-yloxy)-3-fluorophenyl)-4-ethoxy-1-(4-fluorophenyl)-2-oxo-1,2-dihydropyridine-3-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: BMS-777607

INTERVENTIONS:
Drug: BMS-777607 — Suspension/Tablet, Oral, Dose escalation to an MTD from a starting dose of 10 mg, once daily, until disease progression/subject discontinuation

SUMMARY:
Part A: The purpose of this study is to find the maximum tolerated dose of BMS-777607 in subjects with advanced or metastatic solid tumors

Part B: The purpose of this study is to describe the preliminary activity of BMS-77607 in subjects with advanced or metastatic gastroesophageal cancer, hormone refractory prostate cancer, head and neck squamous cell carcinoma, and type I papillary renal cell carcinoma

ELIGIBILITY:
Inclusion Criteria:

Part A:

* Subjects with advanced or metastatic solid tumors who have either progressed on standard therapy or for whom standard therapy is not known

Part B:

* Subjects with advanced or metastatic gastroesophageal cancer, HRPrC, HNSCC, or PRCC who have either progressed on standard therapy, or for whom standard therapy is not known. Eighteen (18) subjects each with gastroesophageal cancer, HRPrC, and HNSCC will be treated. Subjects with PRCC (up to 18) will be enrolled as feasible
* Tumor paraffin tissue block or 6-10 unstained slides from the tumor tissue block must be provided
* Subjects with HRPrC must have either measurable disease or rising PSA levels (≥3 consecutive rising levels with at least 1 week interval and with PSA level ≥5 mg/ml). All other subjects must have measurable disease as assessed by CT or MRI

Exclusion Criteria:

* Know brain metastases
* Uncontrolled or significant cardiovascular disease
* Retinal atrophy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy assessment including vitals signs, physical assessments, and blood tests | will be conducted weekly for the first 3 weeks then every 3 weeks. All assessments will continue for at least 24 months
Tumor assessments | will be conducted every 6 weeks. All assessments will continue for at least 24 months

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of BMS-777607 and its N-oxide metabolite, BMS-797669 | will be assessed once weekly for the first 3 weeks
The effects of BMS-777607 on blood pressure (BP), heart rate (HR) | will be assessed once weekly for the first 3 weeks then every 3 weeks
Effects on electrocardiogram (ECG), PR interval | will be assessed at base line, at week 3 and at end of treatment
Effects on left ventricular function | will be assessed at baseline and every 3 weeks for 1st 6 weeks then once every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- Australia (2):
  - Local Institution, Camperdown, New South Wales
  - Local Institution, Kogarah, New South Wales

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx